CLINICAL TRIAL: NCT06719557
Title: A Two-Part Study to Evaluate the Effects of Multiple Doses of Itraconazole and Multiple Doses of Phenytoin on the Single-Dose Pharmacokinetics of MK-1084 in Healthy Adult Participants
Brief Title: A Study of the Effect of Itraconazole and Phenytoin on Calderasib (MK-1084) in Healthy Adults (MK-1084-008)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 1084-008; MK-1084-008 (Other: MSD); CA43207 (Other: Celerion)
Record Dates: First submitted 2024-12-02; First posted 2024-12-06 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Healthy
MeSH Terms: interventions — Itraconazole; Phenytoin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1: Calderasib + Itraconazole (Experimental): Part 1: In Period 1 participants receive a single dose of calderasib on Day 1 under fasting conditions. In Period 2 participants receive itraconazole once daily (QD) for 7 consecutive days (Day 1 - Day 7), plus a single dose of calderasib administered approximately 2 hours after itraconazole dosing on Day 5. There will be a washout of at least 7 days between dosing in Period 1 and the first dose in Period 2.
  Interventions: Drug: Calderasib; Drug: Itraconazole
- Part 2: Calderasib + Phenytoin (Experimental): Part 2: In Period 1 participants receive a single dose of calderasib on Day 1 under fasting conditions. In Period 2 participants receive phenytoin three times daily (TID) for 14 consecutive days (Day 1 - Day 14), plus a single dose of calderasib co-administered on the morning of Day 13. There will be a washout of at least 7 days between dosing in Period 1 and the first dose in Period 2.
  Interventions: Drug: Calderasib; Drug: Phenytoin

INTERVENTIONS:
Drug: Calderasib — Oral Tablet
  Other Names: MK-1084
Drug: Itraconazole — Oral solution
  Arms: Part 1: Calderasib + Itraconazole
Drug: Phenytoin — Oral capsule (extended)
  Arms: Part 2: Calderasib + Phenytoin

SUMMARY:
The goal of this study is to learn what happens to calderasib in a healthy person's body over time, called a pharmacokinetic (PK) study. Researchers want to compare the amount of calderasib when it is taken as a single dose; with multiple doses of itraconazole, or with multiple doses of phenytoin.

ELIGIBILITY:
Inclusion Criteria:

The main inclusion criteria include but are not limited to the following:

- Has body mass index (BMI) ≥18 kg/m^2 and ≤32 kg/m^2

Exclusion Criteria:

The main exclusion criteria include but are not limited to the following:

* History of cancer (malignancy)
* Positive results for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C virus (HCV)

Part 1 Only:

- History or presence of ventricular dysfunction or risk factors for Torsades de Pointes (e.g., heart failure, cardiomyopathy, family history of Long QT Syndrome)

Pat 2 Only:

- History of seizure (excluding simple febrile seizure), epilepsy, severe head injury, multiple sclerosis, or other known neurological conditions

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2024-05-20 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
Area Under the Concentration-Time Curve from Time 0 to Infinity After Single Dosing (AUC0-Inf) of Calderasib | Pre-dose and at designated time points up to 72 hours post dose
  Blood samples will be collected to determine the AUC0-Inf of calderasib.

SECONDARY OUTCOMES:
Area Under the Concentration-Time Curve from Time 0 to Last Quantifiable Sample (AUC0-last) of Calderasib | Pre-dose and at designated time points up to 72 hours post dose
  Blood samples will be collected to determine the AUC0-last of calderasib.
Area Under the Concentration-Time Curve from Time 0 to 24 hours (AUC0-24) of Calderasib | Pre-dose and at designated time points up to 24 hours post dose
  Blood samples will be collected to determine the AUC0-24 of calderasib.
Maximum Plasma Concentration (Cmax) of Calderasib | Pre-dose and at designated time points up to 72 hours post dose
  Blood samples will be collected to determine the Cmax of calderasib.
Plasma Concentration at 24 Hours (C24) of Calderasib | Pre-dose and at designated time points up to 24 hours post dose
  Blood samples will be collected to determine the C24 of calderasib.
Time to Maximum Plasma Concentration (Tmax) of Calderasib | Pre-dose and at designated time points up to 72 hours post dose
  Blood samples will be collected to determine the Tmax of calderasib.
Apparent Terminal Half-life (t1/2) of Calderasib | Pre-dose and at designated time points up to 72 hours post dose
  Blood samples will be collected to determine the t1/2 of calderasib.
Apparent Clearance (CL/F) of Calderasib | Pre-dose and at designated time points up to 72 hours post dose
  Blood samples will be collected to determine the CL/F of calderasib.
Apparent volume of distribution during terminal phase (Vz/F) of Calderasib | Pre-dose and at designated time points up to 72 hours post dose
  Blood samples will be collected to determine the Vz/F of calderasib.
Number of Participants Who Experience an Adverse Event (AE) | Up to approximately 41 days
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants who experience an AE will be reported.
Number of Participants Who Discontinue Study Treatment Due to an AE | Up to approximately 25 days
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants who discontinue study treatment due to an AE will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (1):
- Celerion (Site 0001), Lincoln, Nebraska, United States

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/